CLINICAL TRIAL: NCT06188637
Title: A Prospective Cell Migration Study in Ulcerative Colitis Patients Treated With Ozanimod (S1P Receptor Antagonist)
Brief Title: Ulcerative Colitis Leukocyte TRAfficking After Treatment With Zeposia: the ULTRAZ Study
Acronym: ULTRAZ
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Funder decision
Sponsor: Geert D'Haens (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Geert D'Haens, Professor, Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-505382-88-00
Record Dates: First submitted 2023-12-15; First posted 2024-01-03 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — ozanimod

STUDY DESIGN:
Intervention Model Description: This is a 2-center prospective open-label study with an 11 week follow-up period and extra disease activity check at week 26.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open- label ozanimod (Experimental): All patients will receive open-label ozanimod
  Interventions: Drug: Ozanimod Oral Capsule

INTERVENTIONS:
Drug: Ozanimod Oral Capsule — open label ozanimod

SUMMARY:
The ULTRAZ study is designed to better understand the mode of action of S1P receptor modulators. The alteration of leukocyte trafficking due to S1P receptors such as ozanimod is mainly investigated in rodent studies. Several previous studies show a reduced total leukocyte count in peripheral blood and only two study reported the effect of leukocyte subgroups before and after treatment with ozanimod. The change in leukocyte subgroups in peripheral blood as well as colonic mucosa and lymph nodes have not been investigated to our knowledge. Therefore, the aim of this study is to explore the changes in these three compartments.

DETAILED DESCRIPTION:
Ozanimod is a sphingosine-1-phosphate (S1P) receptor modulator, which binds with high affinity to receptor subtypes 1 (S1P1) and 5 (S1P5). Many cell types express S1P1, including vascular endothelial cells, brain cells, and leukocytes. Normally, S1P levels are high in blood, heterogeneous in peripheral lymphoid organs (e.g. lymph nodes and Peyer's patches) and low in tissue, creating a gradient. This gradient results in direct trafficking of leukocytes out of the lymph node and into the circulation. In inflamed tissue, increased levels of S1P have been observed, leading to more leukocyte trafficking to this area.

The modulation of the S1P1 receptor by ozanimod causes internalization and desensitization of S1P1 in leukocytes, reducing their migration in response to an increased S1P gradient. Therefore, leukocytes are retained in peripheral lymphoid organs. Previous studies showed a significant - and reversible - reduction of circulating leukocytes in the peripheral blood after treatment with ozanimod, but did not investigate the changes of leukocyte subtypes in colon mucosa and lymphatic system (ie peripheral lymph nodes.

Not all patients respond to treatment with ozanimod. This non-response may be due to a mechanistic failure, where there is ongoing inflammation despite adequate drug concentrations caused by pharmacodynamic failure. The changes in leukocyte subtypes which this study investigates, could give more insight into this type of failure.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-lactating female patients 18 years or older.
2. Documented diagnosis of UC.
3. Active symptomatic UC with endoscopic Mayo score 2-3.
4. Intention to start treatment with ozanimod.
5. Written informed consent.
6. Willing to utilize treatment as prescribed and undergo the procedures that our explained in detail in the informed consent form (ICF).

Exclusion Criteria:

1. Any conditions (e.g., history of alcohol or substance abuse, or lack of compliance) which, in the opinion of the investigator, may interfere with the patient's ability to comply with study procedures.
2. Currently participating, or planning to participate in a study involving an investigational product.
3. Current diagnosis of untreated active tuberculosis, active/chronic hepatitis B. Patients with latent tuberculosis can participate after at least 4 weeks of tuberculostatic treatment per local guidelines.
4. Current gastro-intestinal infection (e.g. C. Diff or other pathogens).
5. Active or planned pregnancy in the year following inclusion.
6. Prior diagnosis of dysplasia in the colon (excluding dysplasia in resected adenomas).
7. History of malignancy in the 5 years prior to randomization except for non-melanoma skin cancer.
8. Abnormal liver function tests and/or abnormal ECG that precludes S1P receptor blocker treatment as per Summary of product characteristics (SmPC).
9. Previous treatment with Vedolizumab (Entyvio).
10. Use of prohibited medication as listed in the SmPC

    -

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
To investigate changes in inflammatory cell subpopulations in the colonic mucosa, the inguinal lymph nodes, and peripheral blood in response to ozanimod induction therapy in patients ulceratie colitis. | Baseline, week 2, 6 and 10.
  To measure the concentration of neutrophils, lymphocytes, monocytes, and dendritic cells at week 0, 2,6 and 10 in the colonic mucosa, the inguinal lymph nodes and peripheral blood using the technique of single cell transcriptomics, spatial transcriptomics and cytometry by time of flight ( CyTOF) in response to ozanimod induction therapy in patients with moderate-to-severe ulcerative colitis.

CONTACTS AND LOCATIONS:
Overall Officials: Geert DHaens, Principal Investigator — AmsterdamUMC

IPD SHARING:
Plan to Share IPD: No